CLINICAL TRIAL: NCT05515146
Title: Lymphovascular Abnormalities Under Tattoos : Preliminary Reports of One Observational Study
Brief Title: Lymphovascular Abnormalities Under Tattoos
Status: Completed | Type: Observational
Sponsor: Haute Ecole Bruxelles-Brabant (Other)
Responsible Party: Principal Investigator, Bourgeois Pierre, Prof Dr P Bourgeois, Haute Ecole Bruxelles-Brabant
Other Study IDs: HE2BHERSICGTT
Record Dates: First submitted 2022-08-15; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Tattoo
Keywords: lymphatic vessels; indocyanin green; near infra red fluorescence lymphatic imaging; tattoo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: near infra red fluorescence lymphatic imaging — ICG (0.2 ml from 25mg of ICG diluted by 5.0 ml of aqua ad injectabilia) was injected intradermally at the basis of the tattooed cutaneous area and at one point chosen so that the tracer had to flow under this area directly towards the root of the limb

SUMMARY:
The number of tattooed people is increasing and some complications secondary to tattoos suggest that the lymphatic vascular system might be implicated in their pathogenesis. Abnormalities have been described at the level of the lymph nodes draining the tattooed areas but nothing was reported about the lymphatic vessels under tattoos. This is the aim of the present work.

DETAILED DESCRIPTION:
19 subjects with 20 tattooed skin surfaces were enrolled after written informed consent and the lymphvascular drainage under the tattooed surface was studied using one near infrared camera device after one intradermal injection of Indocyanine Green.

ELIGIBILITY:
Inclusion Criteria:

* presence of one tattoo at the level of one limb
* written informed consent

Exclusion Criteria:

1. History of iodine allergy or anaphylactic reactions to insect bites or medication;
2. Hyperthyroidism;
3. Severe cardiac or pulmonary disease;
4. Significant renal failure (creatinine > 400 μmol/l);
5. Pregnancy;
6. any known disease of the skin (such as psoriasis);
7. any disease known to affect the cutaneous tissues (such as diabetes);
8. any previous operation and/or trauma at the level of tattooed limb;
9. familial history of lower limb edemas:
10. skin infection after the tattoo

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: nineteen subjects (nine women and ten men; mean age = 28.6, range 23-39 years) with tattoos at the level, either of the lower limb (n = 11), or of the upper limb (n = 9) Except in 4 cases, tattoos were older than 2 years (mean = 52.5 months).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
normal or abnormal lympho-vascular drainage | imagings were performed directly after the injection (duration 3 minutes)
  The following pictures were considered as normal
  - lymphatic vessels are well seen and drainage is fast spontaneously
normal or abnormal lympho-vascular drainage | imagings were performed directly after the stretching and massages (duration 3 minutes)
  The following pictures were considered as normal
  - lymphatic vessels are well seen after stretching and massages of the injected site
normal or abnormal lympho-vascular drainage | imagings were performed after a period of normal activities (duration 30 minutes)
  The following pictures were considered as normal
  - lymphatic vessels are well seen after 30 minutes of normal activities and direct between the injected site and-towards the first lymph node at the root of the limb

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre Bourgeois, Paliseul, Belgium

IPD SHARING:
Plan to Share IPD: No